CLINICAL TRIAL: NCT05925842
Title: Clinical and Molecular Characterization of Axial Psoriatic Arthritis (PsA), A Pilot Study
Acronym: MONOLITH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Group for Research and Assessment of Psoriasis and Psoriatic Arthritis (Network)
Responsible Party: Sponsor
Other Study IDs: MAXPSA001
Record Dates: First submitted 2023-05-10; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with PsA without Axial Involvement
- Participants with PsA with Axial Involvement

SUMMARY:
Objectives: To identify a candidate set of biomarkers specific to AxPsA. Overview: Clinical and imaging characterization of PsA patients will be combined with extensive molecular assessment of both liquid and tissue compartments to identify biomarkers which differentiate PsA patients with and without axial involvement

ELIGIBILITY:
Inclusion Criteria:

* Persons with PsA diagnosed by a consultant Rheumatologist with disease duration of > 3 months but < 10 years with or without IBP.

  * Adults between the ages 18 and 80 years, with joint disease onset after 16 years of age
  * Patients able to understand and complete consent procedures
  * Study participants must have PsA, meet CASPAR criteria, and must have active disease as defined by the treating rheumatologist, including an evaluable psoriatic skin lesion amenable to 6mm punch skin biopsy.

    o Psoriasis should be diagnosed by a consultant rheumatologist or dermatologist.
  * Study participants must have been on consistent therapy for their PsA for the past 90 days
  * Study participants must be naïve to biological treatment and targeted synthetic DMARD treatment (examples: JAK inhibitors, apremilast)

Exclusion Criteria:

* • Persons with musculoskeletal (peripheral or axial) symptoms for >10 years

  * Persons with planned major surgery (e.g., joint replacement) within the duration of the collection of data for the study
  * Persons with a history of chemotherapy, radiation therapy or immunotherapy for cancer in the preceding 5 years.
  * Persons with ongoing cancer (not excluding non-melanoma skin, cervical/breast in-situ carcinoma) but those fully recovered from an episode of cancer (in remission for more than 5 years) may be included at the discretion of the patient's treating rheumatologist.
  * Persons with an active severe or serious infection
  * Patients with non-severe infection at the discretion of the Investigator
  * Persons with other concomitant disorders incompatible with study (at discretion of Investigator).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult persons with diagnosed active PsA including psoriatic lesions, naive to biologic or tsDMARD therapies
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Target biomarker identification | 18 months
  Identify candidate biomarkers able to discriminate between PsA with and without axial involvement

CONTACTS AND LOCATIONS:
Overall Officials: Philip Mease, MD, Principal Investigator — Group for Research and Assessment of Psoriasis and Psoriatic Arthritis; Vinod Chandran, MD, Study Director — Group for Research and Assessment of Psoriasis and Psoriatic Arthritis; Oliver Fitzgerald, MD, Study Director — Group for Research and Assessment of Psoriasis and Psoriatic Arthritis
Locations (2):
- United States (2):
  - University of California San Diego, La Jolla, California
  - Seattle Rheumatology Associates, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No